CLINICAL TRIAL: NCT05616494
Title: A Single-arm, Multicenter, Phase Ⅱ Clinical Study of Docetaxel for Injection (Albumin-bound) in Patients With Pancreatic Cancer Who Have Received at Least One Line of Therapy
Brief Title: A Study of Docetaxel for Injection (Albumin-bound) in Patients With Pancreatic Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HB1801-006
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Docetaxel; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Docetaxel for Injection (Albumin-bound) (Experimental): Docetaxel for Injection (Albumin-bound) will be administrated once every 3 weeks.
  Interventions: Drug: Docetaxel for injection (Albumin-bound)

INTERVENTIONS:
Drug: Docetaxel for injection (Albumin-bound) — Docetaxel for injection (Albumin-bound), by intravenous infusion, every 3 weeks.

SUMMARY:
This trial is a single-arm, multicenter clinical study to evaluate the efficacy and safety of Docetaxel for Injection (Albumin-bound) in patients with pancreatic cancer.

DETAILED DESCRIPTION:
Simon two-stage design will be adopted in this study. In the first stage, 24 patients will be enrolled, if at least 2 of them get response (CR or PR), the second stage of the study will be conducted, and 29 additional patients will be enrolled. If there is only one or no patients get response (CR or PR) in the first stage, the study will be early terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years (subject to the date when the informed consent form is signed) and voluntarily signed the informed consent form.
2. Histologically or cytologically confirmed diagnosis of pancreatic cancer.
3. Patients who have got disease progression or toxic intolerance after previous standard treatment (gemcitabine based and fluorouracil based therapy).
4. At least one measurable lesion according to RECIST v1.1(the measurable lesion area had not received previous radiation therapy or had evidence of definite progression after the end of radiation therapy).
5. Patients with Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
6. Patients with estimated survival time of ≥ 3 months.
7. Patients with fine organ function (no medical supportive treatments such as blood component transfusion, growth factors within 2 weeks before taking the relevant inspections):

   Absolute neutrophil count ≥1.5×10^9/L; Platelets ≥100×10^9/L; Hemoglobin ≥90 g/L; Albumin≥30 g/L; Serum creatinine ≤ 1.5×ULN or creatinine clearance rate ≥ 40 mL/min; Total bilirubin≤1.5 × ULN(≤ 2 × ULN for patients with obstructive jaundice, ≤3 × ULN for patients with Gilbert's syndrome); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3× ULN (≤5× ULN for patients with liver metastasis); Prothrombin time (PT) ≤ 1.5×ULN, International Normalized Ratio (INR) ≤ 1.5×ULN.
8. The patient must agree to take adequate contraception from signing of ICF through 6 months after last dose, women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the first dose of the investigational drug.

Exclusion Criteria:

1. Patients who have a history of severe allergy to any excipients of the investigational drug or taxanes.
2. Patients who had no response to previous taxanes treatments (no tumor shrinkage was observed or disease progressed within 3 months after initiation of the treatment).
3. Patients with partial or complete intestinal obstruction or complete biliary obstruction that cannot be relieved by active treatment.
4. Patients who had a history of other active malignant tumors within 2 years before the first dose of the investigational drug, except for the study disease pancreatic cancer and curable cancer that had been cured (such as basal cell or squamous cell skin cancer, superficial bladder cancer, cervical cancer or breast cancer in situ that had been excised).
5. Patients with brain metastases and meningeal metastases.
6. Patients with chronic hepatitis B (HBsAg and/or HBcAb positive but HBV DNA < 2000 IU/mL can be included), chronic hepatitis C (HCV antibody positive but HCV RNA negative can be included), and HIV antibody positive.
7. Adverse reactions from the previous anti-tumor treatment have not yet recovered to ≤ level 1 based on CTCAE 5.0 (except for alopecia, hyperpigmentation, or other toxicity without safety risk judged by the investigator).
8. Patients with a history of severe cardiovascular disease, including but not limited to:

   1. Severe heart rhythm or conduction abnormalities, including but not limited to ventricular arrhythmia requiring clinical intervention and third degree atrioventricular block within 6 months before the first dose of the investigational drug;
   2. History of myocardial infarction, unstable angina pectoris, angioplasty and coronary artery bypass surgery within 6 months before the first dose of the investigational drug;
   3. Heart failure with New York Heart Association (NYHA) Classification of Class III and above;
   4. Poorly controlled hypertension (Systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg at screening period).
9. Patients with uncontrolled serous cavity effusion requiring frequent drainage or medical intervention (e.g., pleural effusion, abdominal effusion, pericardial effusion, etc., additional intervention was needed within 2 weeks after intervention, excluding exfoliative cytology testing of the exudate) within 7 days before the first dose of the investigational drug.
10. Patients with severe or active infections (including tuberculous infections) that require systemic antibacterial, antifungal, or antiviral therapy within 14 days before the first dose of the investigational drug, antiviral therapy for patients with viral hepatitis is permitted.
11. Patients who have received anti-tumor treatments such as chemotherapy, targeted therapy, immunotherapy and other clinical study drugs within 4 weeks or 5 half-lives of the drugs (whichever is shorter) before the first dose of the investigational drug.
12. Patients who have used potent inhibitors or inducers of CYP3A4 within 2 weeks before the first dose of the investigational drug.
13. Patients who have undergone major surgery within 4 weeks before the first dose of the investigational drug and had not recovered sufficiently, or who need to undergo elective surgery during the study.
14. Pregnant or nursing women.
15. Patients who is participating in another clinical study simultaneously unless it is an observational (non-interventional) clinical study or within the follow-up period of an interventional study.
16. Other situations that the investigator considers not suitable for participating in the clinical study, including but not limited to: the patient is complicated by severe or uncontrolled medical conditions, which will increase the safety risk, interfere with the interpretation of study results or affect the study compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2022-12-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) by Independent Review Committee (IRC) | Up to approximately 2 years

SECONDARY OUTCOMES:
ORR by investigator | Up to approximately 2 years
Overall survival (OS) | Up to approximately 2 years
Disease control rate (DCR) by IRC and investigator | Up to approximately 2 years

OTHER OUTCOMES:
Duration of Response (DoR) by IRC and investigator | Up to approximately 2 years
Progression-Free-Survival (PFS) by IRC and investigator | Up to approximately 2 years
Incidence of AE and SAE | Up to approximately 2 years
Plasma concentration of docetaxel (free and total) | At the end of Cycle 1 (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: xianju Xu, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No